CLINICAL TRIAL: NCT05760703
Title: Phase Ib/II: Multicenter, Open, Dose-escalation Evaluation of the Safety and Efficacy of STSG-0002 Injection in Patients With Chronic Hepatitis B Treated With Oral Antiviral Therapy(Long-term Follow-up)
Brief Title: Evaluate the Safety and Efficacy of STSG-0002 Injection in Patients With Chronic Hepatitis B
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The preliminary effectiveness data observed at present did not meet the expectations, the benefit of the subjects receiving the experimental drug was limited.
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Collaborators: Beijing Sanuo Jiayi Biotechnology Co. LTD (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STS-STSG0002-002-LTFU
Record Dates: First submitted 2023-02-23; First posted 2023-03-08 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- lowest dose treatment group (Experimental): Subjects will receive one single lowest dose of STSG-0002 Injection following protocol requirements
  Interventions: Drug: STSG-0002 Injection
- low dose treatment group (Experimental): Subjects will receive one single low dose of STSG-0002 Injection following protocol requirements
  Interventions: Drug: STSG-0002 Injection
- Intermediate dose treatment group (Experimental): Subjects will receive one single intermediate dose of STSG-0002 Injection following protocol requirements
  Interventions: Drug: STSG-0002 Injection
- A single high dose of treatment group (Experimental): Subjects will receive one single high dose of STSG-0002 Injection following protocol requirements
  Interventions: Drug: STSG-0002 Injection

INTERVENTIONS:
Drug: STSG-0002 Injection — Intravenous infusion

SUMMARY:
This trial is a multi-center, open, single-dose, dose-increasing trial，to evaluate the safety and efficacy of STSG-0002 injection in patients with chronic hepatitis B treated with oral antiviral therapy(Long-term follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic HBV；
* Receiving anti-HB viral therapy；
* 10 IU/ml≤HBsAg≤3000 IU/ml.

Exclusion Criteria:

* Patients co-infected with hepatitis C virus, HIV, HAV, HDV, HEV;
* Liver cirrhosis;
* Hepatocellular carcinoma;
* Autoimmune liver disease;
* Clinical hepatic decompensation;
* Fibroscan>12 kPa;
* a. hemoglobin<110g/L（female）<120 g/L（male），platelet<ULN，white blood cell<2.5×109/L；b. bilirubin>1.5 ×ULN，ALT>2 × ULN，serum albumin<35 g/L；c. INR>1.5；d. serum creatinine >1.5×ULN.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects of adverse events | Baseline to Day 180
Number of subjects With Significant Abnormal Physical Examination | Baseline to Day 180
Number of subjects of Significant Abnormal Vital Signs Findings | Baseline to Day 180
Number of Participants With Significant Abnormal Laboratory Values | Baseline to Day 180
Number of subjects With Significant Abnormal Electrocardiography (ECG) Findings | Baseline to Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, Principal Investigator — Peking University First Hospital
Locations (4):
- China (4):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Youan Hospital,Capital Medical, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No